CLINICAL TRIAL: NCT04705272
Title: The Role of the Living Environment in the Social Inequalities in the Physical Activities of Pregnant Women Residing in the Eurometropole of Strasbourg
Acronym: ENVIFEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7999
Record Dates: First submitted 2020-10-05; First posted 2021-01-12 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Physical Activity of Pregant Women
Keywords: physical activity level; neighborhood,; social inequalities; living environment,; gestational weight gain
MeSH Terms: conditions — Gestational Weight Gain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Pregnant women will be included in the study at the time of their first or second trimester ultrasound in the Hautepierre and CMCO ultrasound department. The period of inclusion should extend from 1 October 2020 to 31 October 2021 with a duration of participation of each subject of 9 months.

SUMMARY:
Excessive weight gain during pregnancy can promote subsequent obesity or increase pre-existing maternal obesity, lead to complications during pregnancy, such as gestational diabetes, hypertension and pre-pregnancy eclampsia, which affect fetal growth.

What are the determinants of excessive weight gain? The first determinant of excessive weight gain is related to healthy living place and physical activity, noted as "PA". Many meta-analyses have demonstrated the role of PA in gestational weight gain.

The main objective is to study the role of the living environment in the PA practice of pregnant women and to identify the socio-environmental construction contributing to the disparities in the practice of PA in women during their pregnancy. This thesis is based on an innovative approach in France, combining both epidemiology and geography approaches to meet priority research objectives in a public health context. With regard to the general issue "What are the contextual determinants of pregnant women's PA practice beyond their individual characteristics that could explain the disparities in practice according to their socio-economic position?" This question underlies the following assumptions:

i) In addition to their individual characteristics, women with low PA and who have reduced PA during pregnancy reside in a more socio-economically deprived neighborhood.

ii)Beyond the socio-economic dimension, the physical characteristic of the residential place influences the level of PA practice of pregnant women.

iii) The combination of the socio-economic, physical and psychosocial environment contributes to reducing the level of PA among pregnant women.

iv) Pregnant women with an unfavourable living environment and low PA have adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women living in the Strasbourg Eurometropolis
* Women performing ultrasound follow-up and giving birth in HUS
* Understanding of the French language
* Patient who has expressed no opposition to the research and/or has signed a consent form in case of collection creation

Exclusion Criteria:

* Refusal to participate in study
* Minor women
* Unable to provide informed information (subject in an emergency, difficulty understanding the subject, etc.)
* Subject under protection of justice
* Subject under guardianship or curatorship
* Obstetric pathologies against-indicating the practice of AP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women will be included in the study at the time of their first or second trimester ultrasound in the Hautepierre and CMCO ultrasound department. The period of inclusion should extend from 1 October 2020 to 31 October 2021 with a duration of participation of each subject of 9 months.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
GWG gestational weight gain | 7 months
  Calculation of the difference in weight at the beginning of pregnancy and at the end of pregnancy based on medical and declarative data

SECONDARY OUTCOMES:
Physical activity during each trimester Pregnancy and delivery outcomes | 7 months
  Measuring physical activity in metabolic equivalents in order to see the progress of this activity

CONTACTS AND LOCATIONS:
Overall Officials: Virginie HAMANN, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Schiltigheim, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simoncic V, Hamann V, Huber L, Deruelle P, Sananes N, Enaux C, Alter M, Schillinger C, Deguen S, Kihal-Talantikite W. Study protocol to explore the social effects of environmental exposure and lifestyle behaviours on pregnancy outcome: an overview of cohort of pregnant women study. BMJ Open. 2022 Sep 17;12(9):e058883. doi: 10.1136/bmjopen-2021-058883. PMID 36115665